CLINICAL TRIAL: NCT02094222
Title: Expanded Access Protocol for an Intermediate Size Population - RAVICTI for Byler Disease
Status: No longer available | Type: Expanded Access
Sponsor: Robert Squires, Jr. (Other)
Responsible Party: Sponsor-Investigator, Robert Squires, Jr., MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO13110219
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Byler Disease
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1 | interventions — glycerol phenylbutyrate

INTERVENTIONS:
Drug: RAVICTI — open label expanded access protocol of titrated dosing regimen of RAVICTI for up to 60 weeks
  Other Names: glycerol phenylbutyrate

SUMMARY:
Byler Disease is the result of a homozygous missense (G308V) mutation in the ATP8B1 gene. The disease is typically manifest in the first year of life on the basis of complications of cholestasis; common presentations include jaundice, poor growth, bleeding related to vitamin K deficiency, and/or weak bones related to vitamin D deficiency. Early management of Byler Disease is directed at nutritional issues which tend to be responsive to medical intervention, unlike the pruritus/scratching which remains a devastating problem. Progressive liver disease develops in Byler Disease and can lead to cirrhosis and end-stage liver disease. This is an open label expanded access protocol of RAVICTI in children with Byler Disease. The primary hypothesis is that the administration of RAVICTI in these children is feasible, well tolerated and safe. It is also hypothesized that RAVICTI treatment leads to an improvement in biochemical markers of liver disease and it may ameliorates or prevents the development of scratching behavior as a manifestation of pruritus attributed to the liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Byler Disease as identified by a homozygous mutation in ATP8B1 predicted to yield a G308V missense mutation
* Total serum bile acid > 100 µM
* Male or female subjects of age greater than 130 days to begin screening procedures
* Male or female subjects of age greater than 180 days to begin RAVICTI therapy
* Ability and willingness to adhere to all study protocols
* Access to intermittent phone contact
* Written informed consent

Exclusion Criteria:

* Prior surgical interruption of the enterohepatic circulation (including but not limited to partial biliary diversion and/or ileal exclusion)
* Liver transplantation
* Other diagnosed concomitant liver disease
* Evidence of portal hypertension

  * Platelet count < 150,000 and
  * Spleen palpable > 2 cm below the costal margin, or
  * History of a clinical complication/feature c/w portal hypertension
* esophageal or gastric varix or variceal hemorrhage
* ascites
* hepatic encephalopathy
* Coagulopathy (PT > 15 seconds or INR > 1.5) despite vitamin K therapy
* ALT > 10 X ULN
* Allergy/hypersensitivity to RAVICTI or 4-phenylbutyrate
* Severe concurrent illnesses, such as neurological, cardiovascular, pulmonary, metabolic, endocrine, and renal disorders, that would interfere with the conduct and results of the study
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Cancer or history of cancer
* Any female who is pregnant or lactating or who is planning to become pregnant with 1 year of enrollment
* Any known history of alcohol or substance abuse

Ages: 130 Days to 21 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Squires, MD, Principal Investigator — University of Pittsburgh